CLINICAL TRIAL: NCT04393740
Title: The Contribution of Posterior Corneal Astigmatism to Total Corneal Astigmatism Using Scheimpflug Analyzer (Pentacam ) in a Sample of Egyptian Population
Brief Title: Contribution of Posterior Corneal Astigmatism to Total Corneal Astigmatism in a Sample of Egyptian Population
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Mohamed Badawy, Resident of ophthalmology kasr el AINI, Cairo University
Other Study IDs: Ms-184-2019
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Corneal Astigmatism
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: scheimpflug imaging using pentacam — corneal tomography imaging using pentacam device (based on Scheimpflug principle )

SUMMARY:
The magnitude of posterior corneal astigmatism was considered negligible due to the smaller difference in the refractive index between the cornea and the aqueous .

though ,neglecting the posterior corneal astigmatism lead to errors during calculation of the toric iols (over or under estimation ) .

so we aim to determine the percentage of contribution of posterior corneal astigmatism to total corneal astigmatism in a sample of Egyptian population using scheimpflug imaging (Pentacam ).

DETAILED DESCRIPTION:
Astigmatism is a common vision condition that causes blurred vision. Astigmatism is an error of refraction in which incident parallel rays can't be focused to a single point .It could be corneal or lenticular astigmatism or both . Regarding Corneal astigmatism it is due to difference in the corneal curvature in the different meridian of both the anterior and posterior surface .

The are 2 methods of studing corneal curvature :

* Corneal topography which depend on placcido disc to study anterior corneal surface .
* Corneal tomography is more precise in detecting anterior and posterior corneal curvature depending on Scheimpflug principle which uses a rotating Scheimpflug camera .

Pentacam is a device which depend on Scheimpflug technique .

The importance of studing the posterior corneal curvature includes :

• The posterior corneal curvature is a more sensitive indicator of early keratoconus detection especially posterior corneal elevation.

Previously, The change in the posterior corneal surface plays a more subtle role than the anterior corneal surface in optical performance because of the smaller difference in refractive indices between the cornea and aqueous, and it has been thought that the magnitude of PCA in the normal population is clinically negligible.

Posterior corneal astigmatism (PCA) is important for better predictability of toric intraocular lens calculation to avoid under- or overestimation of toricity in intraocular lens (IOL) power calculations.

But recently it has been demonstrated how neglecting PCA will lead to overcorrection of astigmatism in eyes with with-the-rule astigmatism (WTR) and undercorrection in eyes with against-the-rule astigmatism (ATR).(3) In our study we aim to Determine the contribution of posterior corneal astigmatism to total corneal astigmatism and the error in estimating total corneal astigmatism from anterior corneal measurements only using Scheimpflug analyzer (Pentacam ).

Our patients will undergo Scheimpflug imaging using pentacam .

From the corneal parameters displayed in pentacam we can calculate :

* Anterior corneal astigmatism by substracting Ksteep -Kflat on the front surface
* Posterior corneal astigmatism by substracting Ksteep-Kflat on the back surface.
* Total corneal astigmatism is calculated by addition of anterior and posterior corneal astigmatism using vector analysis by using ASSORT vector calculator.*
* The percentage of contribution of posterior corneal astigmatism to magnitude of Total corneal astigmatism is then calculated .

ASSORT vector calculator:

Is a total planning and outcomes analysis software for astigmatism using Alpins method ,cheltman ,Victoria ,Australia .

ELIGIBILITY:
Inclusion Criteria:

1. Patients with corneal astigmatism(±0.5D up tp ±4 D )
2. Age (18-45 years )
3. Refractive error (myopia up to -8D)
4. Hyperopia up to +4
5. Patients who have clear cornea .
6. Good quality Scheimpflug analyzer scans.

Exclusion Criteria:

1. Patients who have any corneal opacity .
2. Patients who underwent any Previous corneal surgery .
3. Patients who have Co existing corneal pathology.
4. Glaucomatus patients.
5. Patients with any Concomitant ocular disease .
6. Patients with History of previous ocular trauma .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: candidates presenting for refractive surgery .
Sampling Method: Non-Probability Sample
Enrollment: 356 (Estimated)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-08-15 (Estimated)

PRIMARY OUTCOMES:
contribution of posterior corneal astigmatism to magnitude of total corneal astigmatism | 3 months
  to detect the contribution of posterior corneal astigmatism to total corneal astigmatism to avoid errors during calculation of toric Intra ocular lenses

CONTACTS AND LOCATIONS:
Locations (1):
- kasr El Aini medical school, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
we would share our protocol and results through publishing our research
Supporting Information: Study Protocol
Time Frame: the data would be available within 3 months and would be available for 6 months

REFERENCES:
- [Background] Ferreira TB, Ribeiro P, Ribeiro FJ, O'Neill JG. Comparison of Methodologies Using Estimated or Measured Values of Total Corneal Astigmatism for Toric Intraocular Lens Power Calculation. J Refract Surg. 2017 Dec 1;33(12):794-800. doi: 10.3928/1081597X-20171004-03. PMID 29227506
- [Background] Rydstrom E, Westin O, Koskela T, Behndig A. Posterior corneal astigmatism in refractive lens exchange surgery. Acta Ophthalmol. 2016 May;94(3):295-300. doi: 10.1111/aos.12965. Epub 2016 Jan 30. PMID 26825986